CLINICAL TRIAL: NCT01090388
Title: A Cross-Sectional Study Of Patient-Reported Outcomes For Bladder Cancer Patients With Non-Invasive Disease
Brief Title: Bladder Cancer Patient-Reported Outcomes
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, David Latini, Associate Professor of Urology, Baylor College of Medicine
Other Study IDs: SDU07-BlCa-PRO
Record Dates: First submitted 2008-07-16; First posted 2010-03-22 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Bladder Neoplasms
Keywords: Cross-sectional survey; Health-related quality of life; Symptom management
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Participants voluntarily completed a telephone interview using a questionnaire compiled using validated, patient-centered measures of cancer outcomes and psychosocial status.

SUMMARY:
The purpose of this study is to identify aspects of the bladder cancer (BlCa) survivorship experience that differ by clinical risk at diagnosis. The investigators will collect cross-sectional data from persons with BlCa to identify aspects of health-related quality of life (HRQOL) and symptom management. The study originally enrolled only nonmuscle-invasive bladder cancer survivors but has been expanded to include survivors with any stage disease. Information from this study will be used to develop a new patient education and counseling intervention.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Diagnosed with BlCa within the past 4 years
* Able to read, speak, and understand English
* Able to provide informed consent.

Exclusion Criteria:

* Younger than 18
* Diagnosed BlCa longer than 4 years ago
* Unable to read, speak, and understand English
* Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bladder cancer patients (all stages) recruited at hospitals affiliated with Baylor College of Medicine and MD Anderson Cancer Center and via the websites of bladder cancer survivor organizations
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2007-07; Primary Completion 2011-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life as measured by the EORTC QLQ C30 and BLS24 (nonmuscle-invasive) or BLM30 (muscle-invasive or metastatic) | Duration of Study
  Health-related quality of life as measured by the European Organization for Resarch and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30 and BLS24 (that is, BLadder cancer Superficial, meaning nonmuscle-invasive) or BLM30 (BLadder cancer muscle-invasive or metastatic).
  Data are assessed at one time point only. Survey participants may be assessed at any point between diagnosis and 4 years post-diagnosis. The questions in the survey typically ask about health-related quality of life in the preceding 4 weeks.

SECONDARY OUTCOMES:
Illness intrusiveness | Duration of Study
  Data are assessed at one time point only. Survey participants may be assessed at any point between diagnosis and 4 years post-diagnosis. The questions in the survey typically ask about health-related quality of life in the preceding 4 weeks.
CaPSURE Fear of Recurrence | Duration of Study
  The fear of recurrence measure was originally developed and validated for the Cancer of the Prostate Strategic Urologic Research Endeavor (CaPSURE) study.
  Data are assessed at one time point only. Survey participants may be assessed at any point between diagnosis and 4 years post-diagnosis. The questions in the survey typically ask about health-related quality of life in the preceding 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: David M Latini, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Background] Latini DM, Lerner SP, Wade SW, Lee DW, Quale DZ. Bladder cancer detection, treatment and outcomes: opportunities and challenges. Urology. 2010 Feb;75(2):334-9. doi: 10.1016/j.urology.2009.09.051. Epub 2009 Dec 5. PMID 19963252
- [Result] Kowalkowski MA, Chandrashekar A, Amiel GE, Lerner SP, Wittmann DA, Latini DM, Goltz HH. Examining sexual dysfunction in non-muscle-invasive bladder cancer: results of cross-sectional mixed-methods research. Sex Med. 2014 Aug;2(3):141-51. doi: 10.1002/sm2.24. PMID 25356311
- [Result] Kowalkowski MA, Goltz HH, Petersen NJ, Amiel GE, Lerner SP, Latini DM. Educational opportunities in bladder cancer: increasing cystoscopic adherence and the availability of smoking-cessation programs. J Cancer Educ. 2014 Dec;29(4):739-45. doi: 10.1007/s13187-014-0649-3. PMID 24719024